CLINICAL TRIAL: NCT05532007
Title: Effects of Peanut Intake on Task-related Brain Activation and Cognitive Functions in Older Adults With Memory Complaints: A Randomized Controlled Study
Brief Title: Effects of Peanut Intake on Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: The Peanut Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5210436
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cognition; Inflammation
Keywords: Peanuts; cognition; inflammation; oxidative stress
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This is a free living , randomized, controlled, parallel design study with 30 subjects, who will be randomized to either receive peanuts or abstain from them for 12 weeks.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participants will be aware if they received the intervention or not, however, the cognitive testers and FMRI techs would not be aware of the participant randomization group and neither will the data analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut Group (Active Comparator): Peanuts: 2-3 ounces per day to replace 20% of daily energy intake
  Interventions: Dietary Supplement: Peanuts
- Control Group (Active Comparator): Habitual diet abstain from eating peanuts
  Interventions: Other: Habitual Diet

INTERVENTIONS:
Dietary Supplement: Peanuts — 2-3 ounces of peanuts to replace 20% of total daily energy intake
  Arms: Peanut Group
Other: Habitual Diet — continue with habitual diet and abstain from eating peanuts
  Arms: Control Group

SUMMARY:
The study will test the effects of Peanuts on task-related brain activation and cognitive functions in older adults with memory complaints.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of peanuts on cognitive performance and task-related brain activation on functional magnetic resonance imaging (fMRI) in older adults. The specific aim of the study is to explore the neuroprotective effects of a peanut-enriched diet (2-3 oz of peanuts to replace 20% of the total energy of the habitual diet) for 12 weeks compared to a peanut-excluded habitual diet in elderly men and women with increased risk for CVD and self-reported memory complaints. The study population is older adults 60-80 years in age.

ELIGIBILITY:
Inclusion Criteria:

* Non-demented elderly between 60-80 years of age
* Self-reported memory complaints
* Two cardiovascular risk factors
* Stable weight for at least 6 months prior to recruitment

Exclusion Criteria:

* Peanut allergy
* Smoker
* Endocrine, metabolic and neuropsychological disorders
* Ineligible to get an MRI
* Consuming more than 3 servings/week of nuts including peanuts

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
changes from baseline in Brian activation | baseline to 12 weeks
  Changes will be assessed by Functional MRI (fMRI) on participants. there is no units of measure
changes from baseline serum markers of inflammation | baseline to 12 weeks
  changes in serum inflammation markers which includes hs-CRP, IL-6, TNF-α, ICAM/VCAM, eSelectin, F2-isoprostanes, 8-hydroxy-deoxyguanosine (8-OH-dG) will all be assessed using ELISA

SECONDARY OUTCOMES:
changes from baseline in global cognitive composite score | baseline to 12 weeks
  The composite score will be calculated using the scores from the tests listed below. We will calculate the standardized scores of each test as the score of each participant minus the group mean and divide by its standard deviation. The composite score is the mean of the standardized scores. the 5 tests are: Rey Auditory Verbal Learning Test (RAVLT), Brief Visuospatial Memory Test, Digit Span, FAS Word Fluency, Symbol Digit Modalities Test
Change in serum brain-derived neurotrophic factor (pg/mL) | baseline to 12 weeks
  changes in serum brain-derived neurotrophic factor (pg/mL) assessed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Sujatha Rajaram, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States